CLINICAL TRIAL: NCT05722275
Title: Prediction of Peritoneal Metastasis for Gastric Cancer Based on Radiomics: a Multi-center Prospective Study
Brief Title: Prediction of Peritoneal Metastasis for Gastric Cancer Based on Radiomics
Status: Recruiting | Type: Observational
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: Peking University Cancer Hospital & Institute (Other); Zhenjiang First People's Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Nanfang Hospital, Southern Medical University (Other); Guizhou Provincial People's Hospital (Other); Henan Cancer Hospital (Other Government); Yunnan Cancer Hospital (Other); Guangdong Provincial People's Hospital (Other); Guangzhou Medical University (Other); Fujian Medical University Union Hospital (Other); Shanxi Province Cancer Hospital (Other); Sun Yat-sen University (Other); Beihang University (Other); Scientific Institute San Raffaele (Other)
Responsible Party: Principal Investigator, Di Dong, Professor, Chinese Academy of Sciences
Other Study IDs: CASMI003
Record Dates: First submitted 2022-12-30; First posted 2023-02-10 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Gastric Cancer; Peritoneal Metastases
Keywords: Artificial Intelligence; Classification; Gastric Cancer; Peritoneal Metastases; Computed Tomography; Radiomics
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (13):
- Peking University Cancer Hospital & Institute: Peking University Cancer Hospital & Institute collects clinical information, preoperative CT images, and the golden standard for peritoneal metastasis status for each patient. Clinical information includes gender, age, gastric disease background, tumor markers, gastric cancer stage, gastric cancer type, treatment program, smoking history, alcohol history, etc. All patients undergo diagnostic laparoscopy. Any suspicious lesion discovered during laparoscopy is biopsied and pathologically examined to determine peritoneal metastasis status.
  Interventions: Diagnostic Test: Peritoneal metastasis status ascertainment
- Zhenjiang First People's Hospital: Zhenjiang First People's Hospital collects clinical information, preoperative CT images, and the golden standard for peritoneal metastasis status for each patient. Clinical information includes gender, age, gastric disease background, tumor markers, gastric cancer stage, gastric cancer type, treatment program, smoking history, alcohol history, etc. All patients undergo diagnostic laparoscopy. Any suspicious lesion discovered during laparoscopy is biopsied and pathologically examined to determine peritoneal metastasis status.
  Interventions: Diagnostic Test: Peritoneal metastasis status ascertainment
- The First Affiliated Hospital of Zhengzhou University: The First Affiliated Hospital of Zhengzhou University collects clinical information, preoperative CT images, and the golden standard for peritoneal metastasis status for each patient. Clinical information includes gender, age, gastric disease background, tumor markers, gastric cancer stage, gastric cancer type, treatment program, smoking history, alcohol history, etc. All patients undergo diagnostic laparoscopy. Any suspicious lesion discovered during laparoscopy is biopsied and pathologically examined to determine peritoneal metastasis status.
  Interventions: Diagnostic Test: Peritoneal metastasis status ascertainment
- Nanfang Hospital of Southern Medical University: Nanfang Hospital of Southern Medical University collects clinical information, preoperative CT images, and the golden standard for peritoneal metastasis status for each patient. Clinical information includes gender, age, gastric disease background, tumor markers, gastric cancer stage, gastric cancer type, treatment program, smoking history, alcohol history, etc. All patients undergo diagnostic laparoscopy. Any suspicious lesion discovered during laparoscopy is biopsied and pathologically examined to determine peritoneal metastasis status.
  Interventions: Diagnostic Test: Peritoneal metastasis status ascertainment
- Guizhou Provincial People's Hospital: Guizhou Provincial People's Hospital collects clinical information, preoperative CT images, and the golden standard for peritoneal metastasis status for each patient. Clinical information includes gender, age, gastric disease background, tumor markers, gastric cancer stage, gastric cancer type, treatment program, smoking history, alcohol history, etc. All patients undergo diagnostic laparoscopy. Any suspicious lesion discovered during laparoscopy is biopsied and pathologically examined to determine peritoneal metastasis status.
  Interventions: Diagnostic Test: Peritoneal metastasis status ascertainment
- Henan Cancer Hospital: Henan Cancer Hospital collects clinical information, preoperative CT images, and the golden standard for peritoneal metastasis status for each patient. Clinical information includes gender, age, gastric disease background, tumor markers, gastric cancer stage, gastric cancer type, treatment program, smoking history, alcohol history, etc. All patients undergo diagnostic laparoscopy. Any suspicious lesion discovered during laparoscopy is biopsied and pathologically examined to determine peritoneal metastasis status.
  Interventions: Diagnostic Test: Peritoneal metastasis status ascertainment
- Yunnan Cancer Hospital: Yunnan Cancer Hospital collects clinical information, preoperative CT images, and the golden standard for peritoneal metastasis status for each patient. Clinical information includes gender, age, gastric disease background, tumor markers, gastric cancer stage, gastric cancer type, treatment program, smoking history, alcohol history, etc. All patients undergo diagnostic laparoscopy. Any suspicious lesion discovered during laparoscopy is biopsied and pathologically examined to determine peritoneal metastasis status.
  Interventions: Diagnostic Test: Peritoneal metastasis status ascertainment
- Guangdong Provincial People's Hospital: Guangdong Provincial People's Hospital collects clinical information, preoperative CT images, and the golden standard for peritoneal metastasis status for each patient. Clinical information includes gender, age, gastric disease background, tumor markers, gastric cancer stage, gastric cancer type, treatment program, smoking history, alcohol history, etc. All patients undergo diagnostic laparoscopy. Any suspicious lesion discovered during laparoscopy is biopsied and pathologically examined to determine peritoneal metastasis status.
  Interventions: Diagnostic Test: Peritoneal metastasis status ascertainment
- Guangzhou Medical University: Affiliated Cancer Hospital and Institute of Guangzhou Medical University collects clinical information, preoperative CT images, and the golden standard for peritoneal metastasis status for each patient. Clinical information includes gender, age, gastric disease background, tumor markers, gastric cancer stage, gastric cancer type, treatment program, smoking history, alcohol history, etc. All patients undergo diagnostic laparoscopy. Any suspicious lesion discovered during laparoscopy is biopsied and pathologically examined to determine peritoneal metastasis status.
  Interventions: Diagnostic Test: Peritoneal metastasis status ascertainment
- Fujian Medical University Union Hospital: Fujian Medical University Union Hospital collects clinical information, preoperative CT images, and the golden standard for peritoneal metastasis status for each patient. Clinical information includes gender, age, gastric disease background, tumor markers, gastric cancer stage, gastric cancer type, treatment program, smoking history, alcohol history, etc. All patients undergo diagnostic laparoscopy. Any suspicious lesion discovered during laparoscopy is biopsied and pathologically examined to determine peritoneal metastasis status.
  Interventions: Diagnostic Test: Peritoneal metastasis status ascertainment
- Shanxi Province Cancer Hospital: Shanxi Province Cancer Hospital collects clinical information, preoperative CT images, and the golden standard for peritoneal metastasis status for each patient. Clinical information includes gender, age, gastric disease background, tumor markers, gastric cancer stage, gastric cancer type, treatment program, smoking history, alcohol history, etc. All patients undergo diagnostic laparoscopy. Any suspicious lesion discovered during laparoscopy is biopsied and pathologically examined to determine peritoneal metastasis status.
  Interventions: Diagnostic Test: Peritoneal metastasis status ascertainment
- Sun Yat-sen University: Sun Yat-sen University collects clinical information, preoperative CT images, and the golden standard for peritoneal metastasis status for each patient. Clinical information includes gender, age, gastric disease background, tumor markers, gastric cancer stage, gastric cancer type, treatment program, smoking history, alcohol history, etc. All patients undergo diagnostic laparoscopy. Any suspicious lesion discovered during laparoscopy is biopsied and pathologically examined to determine peritoneal metastasis status.
  Interventions: Diagnostic Test: Peritoneal metastasis status ascertainment
- Scientific Institute San Raffaele: Scientific Institute San Raffaele collects clinical information, preoperative CT images, and the golden standard for peritoneal metastasis status for each patient. Clinical information includes gender, age, gastric disease background, tumor markers, gastric cancer stage, gastric cancer type, treatment program, smoking history, alcohol history, etc. All patients undergo diagnostic laparoscopy. Any suspicious lesion discovered during laparoscopy is biopsied and pathologically examined to determine peritoneal metastasis status.
  Interventions: Diagnostic Test: Peritoneal metastasis status ascertainment

INTERVENTIONS:
Diagnostic Test: Peritoneal metastasis status ascertainment — Each participant with gastric cancer will undergo enhanced CT examination for detection of peritoneal metastasis. Within two weeks of CT examination, the participant will undergo diagnostic laparoscopy to confirm the status of peritoneal metastasis.

SUMMARY:
Peritoneal metastasis of gastric cancer is difficult to be detected in time, thus delaying treatment. Based on the conventional CT images of gastric cancer, this study plans to develop, improve and validate an intelligent analysis system based on radiomics. By extracting and combining the radiomics features related to peritoneal metastasis of gastric cancer, the intelligent analysis system could predict the risk of peritoneal metastasis, and provide personalized decision suggestions for the treatment of gastric cancer.

DETAILED DESCRIPTION:
Peritoneal metastasis of gastric cancer is difficult to be detected in time, thus delaying treatment. Based on the conventional CT images of gastric cancer, this study plans to develop, improve and validate an intelligent analysis system based on radiomics. By extracting and combining the radiomics features related to peritoneal metastasis of gastric cancer, the intelligent analysis system could predict the risk of peritoneal metastasis, and provide personalized decision suggestions for the treatment of gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* (1) diagnosed advanced gastric cancer (≥cT3) by endoscopy-biopsy pathology, combined with CT and/or endoscopic ultrasound;
* (2) with both enhanced CT and laparoscopy;
* (3) without typical peritoneal metastasis indications in CT (diffuse omental nodules or omental cake, large amount of ascites, obvious irregular thickening with high peritoneal enhancement);
* (4) without other evidence of distant metastasis, and no stage IV features on CT.

Exclusion Criteria:

* (1) previous abdominal surgery;
* (2) previous abdominal malignancies or inflammatory diseases;
* (3) time intervals between CT and laparoscopy longer than 2 weeks;
* (4) CT image artifacts that undermine peritoneal lesion assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All included patients are initially diagnosed as peritoneal metastasis-negative by CT, but later confirmed with the actual peritoneal metastasis status in laparoscopic exploration.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The aera under the receiver operating characteristic curve (AUC) of intelligent analysis system | three months
  AUC of the intelligent analysis system in predicting peritoneal metastasis for gastric cancer.

SECONDARY OUTCOMES:
The accuray of intelligent analysis system in predicting peritoneal metastasis | three months
  The agreement between the prediction outcome of intelligent analysis system and the golden standard of peritoneal metastasis.

OTHER OUTCOMES:
The statistical significance of intelligent analysis system in risk stratification | Three years
  Statistical significance (P value) of progression-free survival (PFS) in gastric cancer patients between high-risk and low-risk group identified by the intelligent analysis system.
Progression-free survival time | Three years
  The progression-free survival time in patient subgroups stratified by the intelligent analysis system.
Overall survival | Three years
  The overall survival time in patient subgroups stratified by the intelligent analysis system.

CONTACTS AND LOCATIONS:
Locations (13):
- China (12):
  - Peking University Cancer Hospital & Institute, Beijing
  - Fujian Medical University Union Hospital, Fuzhou
  - Affiliated Cancer Hospital and Institute of Guangzhou Medical University, Guangzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - Nanfang Hospital of Southern Medical University, Guangzhou
  - Sun Yat-Sen University Cancer Hospital, Guangzhou
  - Guizhou Provincial People's Hospital, Guiyang
  - Yunnan Cancer Hospital, Kunming
  - Shanxi Province Cancer Hospital, Taiyuan
  - Henan Cancer Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Zhenjiang First People's Hospital, Zhenjiang
- Scientific Institute San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Smyth EC, Verheij M, Allum W, Cunningham D, Cervantes A, Arnold D; ESMO Guidelines Committee. Gastric cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2016 Sep;27(suppl 5):v38-v49. doi: 10.1093/annonc/mdw350. No abstract available. PMID 27664260
- [Background] Ajani JA, D'Amico TA, Bentrem DJ, Chao J, Cooke D, Corvera C, Das P, Enzinger PC, Enzler T, Fanta P, Farjah F, Gerdes H, Gibson MK, Hochwald S, Hofstetter WL, Ilson DH, Keswani RN, Kim S, Kleinberg LR, Klempner SJ, Lacy J, Ly QP, Matkowskyj KA, McNamara M, Mulcahy MF, Outlaw D, Park H, Perry KA, Pimiento J, Poultsides GA, Reznik S, Roses RE, Strong VE, Su S, Wang HL, Wiesner G, Willett CG, Yakoub D, Yoon H, McMillian N, Pluchino LA. Gastric Cancer, Version 2.2022, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2022 Feb;20(2):167-192. doi: 10.6004/jnccn.2022.0008. PMID 35130500
- [Background] Hur H, Lee HH, Jung H, Song KY, Jeon HM, Park CH. Predicting factors of unexpected peritoneal seeding in locally advanced gastric cancer: indications for staging laparoscopy. J Surg Oncol. 2010 Dec 1;102(7):753-7. doi: 10.1002/jso.21685. PMID 20812349
- [Background] Burbidge S, Mahady K, Naik K. The role of CT and staging laparoscopy in the staging of gastric cancer. Clin Radiol. 2013 Mar;68(3):251-5. doi: 10.1016/j.crad.2012.07.015. Epub 2012 Sep 14. PMID 22985749
- [Result] Dong D, Tang L, Li ZY, Fang MJ, Gao JB, Shan XH, Ying XJ, Sun YS, Fu J, Wang XX, Li LM, Li ZH, Zhang DF, Zhang Y, Li ZM, Shan F, Bu ZD, Tian J, Ji JF. Development and validation of an individualized nomogram to identify occult peritoneal metastasis in patients with advanced gastric cancer. Ann Oncol. 2019 Mar 1;30(3):431-438. doi: 10.1093/annonc/mdz001. PMID 30689702